CLINICAL TRIAL: NCT00002366
Title: A Phase II Safety and Activity Study of Ritonavir in the Treatment of HIV-Associated Cutaneous Kaposi's Sarcoma
Brief Title: The Safety and Effectiveness of Ritonavir in the Treatment of HIV-Related Kaposi's Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott (Industry)
Purpose: Treatment
Other Study IDs: 245C; M95-320
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2009-02-20 (Estimated); Status verified 2009-02

CONDITIONS: Sarcoma, Kaposi; HIV Infections
Keywords: Skin Neoplasms; Sarcoma, Kaposi; Acquired Immunodeficiency Syndrome; HIV Protease Inhibitors; Ritonavir
MeSH Terms: conditions — Sarcoma, Kaposi; HIV Infections; Skin Neoplasms; Acquired Immunodeficiency Syndrome | interventions — Ritonavir

INTERVENTIONS:
Drug: Ritonavir

SUMMARY:
To evaluate the safety and anti-Kaposi's sarcoma activity of ritonavir.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Patients may receive oral acyclovir and may continue prophylactic treatment for PCP, fungal infection, MAC and toxoplasmosis.
* Topical treatment and intralesional chemotherapy will be allowed for lesions which will not be used as indicator or biopsy lesions.

Concurrent Treatment:

Allowed:

Localized radiotherapy will be allowed for lesions which will not be used as indicator or biopsy lesions.

Patients must have:

* Documentation of a positive ELISA test for HIV with a confirmatory test.
* Biopsy proven, cutaneous or oropharyngeal Kaposi's sarcoma.
* Vital signs, physical examination and laboratory assessments that exhibit no evidence of an acute illness.
* Patients must agree to report all current medications to the primary investigator and obtain prior permission to use them when feasible.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms and conditions are excluded:

* Evidence of pulmonary Kaposi's sarcoma.
* Positive urine screen for recreational drugs.
* Current participation in another antiviral research study.
* Investigator anticipates poor patient compliance with the protocol.
* Patient has any condition that, in the investigator's opinion, may obscure the proper observation of the safety or activity of ritonavir.

Concurrent Medication:

Excluded:

* Antiretroviral therapy.
* Protease inhibitor therapy.
* Antiviral agent (e.g., oral ganciclovir or Foscarnet) or prophylactic medication for an AIDS defining illness which the patient cannot be removed from.
* Chemotherapy for Kaposi's sarcoma.
* Treatment with any medications that may interact with ritonavir.

Concurrent Treatment:

Excluded:

Radiotherapy for Kaposi's sarcoma.

Patients with any of the following prior conditions are excluded:

* History of psychiatric illness which is currently medically significant.
* History of pancreatitis.

Prior Medication:

Excluded:

* All antiretroviral therapy within 2 weeks prior to the start of the treatment phase of the study.
* Systemic chemotherapy of interferon within 30 days prior to study entry.
* Previous treatment with a protease inhibitor.

Risk Behavior:

Excluded:

Active substance abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - Prince Henry's Hosp / Med Oncology, Sydney
  - Saint Vincent's Hosp Med Centre, Sydney

REFERENCES:
- [Background] Carr A, Milliken S, Lewis C, Mitsuyasu R, Miles S, Newell M, Cooper DA. A pilot phase II safety and activity study of ritonavir in the treatment of HIV-associated cutaneous Kaposi's sarcoma. Conf Retroviruses Opportunistic Infect. 1997 Jan 22-26;4th:194 (abstract no 703)